CLINICAL TRIAL: NCT02287935
Title: Effectiveness of Limberg and Karydakis Flap in Recurrent Pilonidal Sinus Disease
Brief Title: Limberg and Karydakis Flap in Recurrent Pilonidal Sinus Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adana Numune Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Aziret, Doc. Dr. Selim Sözen, A. Prof. Dr. İlhan Bali, Adana Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AdanaNTRH
Record Dates: First submitted 2014-10-24; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Recurrent Pilonidal Sinus Disease
Keywords: Karydakis procedure; Limberg flap; recurrent pilonidal sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Limberg flap (Active Comparator): Patients were divided into two groups, group 1 were treated with Limberg flap technique
  Interventions: Procedure: Limberg flap
- Karydakis procedure (Active Comparator): Patients were divided into two groups, group 2 were treated with Karydakis procedure
  Interventions: Procedure: Karydakis procedure

INTERVENTIONS:
Procedure: Limberg flap — Patients were divided into two groups, group 1 were treated with Limberg flap technique (n= 37) . Two groups were compared with a statistical in terms of fluid collection, wound infection, flap edema, hematoma, partial wound separation, return to daily activities, pain score, completes healing time, painless seating and patient satisfactions
  Arms: Limberg flap
Procedure: Karydakis procedure — Patients were divided into two groups, group 2 were treated with Karydakis flap (n= 34). Two groups were compared with a statistical in terms of fluid collection, wound infection, flap edema, hematoma, partial wound separation, return to daily activities, pain score, completes healing time, painless seating and patient satisfactions
  Arms: Karydakis procedure

SUMMARY:
It was investigated whether there is a factor that can aid determination of the preferred technique by comparing the early Limberg flap and Karydakis procedure techniques for the treatment of recurrent pilonidal sinus.

DETAILED DESCRIPTION:
Sacrococcygeal pilonidal sinus is common in young men and may recur overtime after surgery.

It was investigated whether there is a factor that can aid determination of the preferred technique by comparing the early Limberg flap and Karydakis procedure techniques for the treatment of recurrent pilonidal sinus.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to give written informed consent
2. There should be recurrent pilonidal sinus

2. Recurrent adult patients (over 18 years of age) undergoing surgery for pilonidal sinus

3. International normalizing ratio (INR) less than 1.5

4. Prothrombin time (PT) should be less than 15 s

5. Partial thromboplastin (PTT) time should be near normal

6. Platelet count should be greater than 50,000 per mm3 to limit the risk of bleeding

7. There must be no infection at the time of surgery

-

Exclusion Criteria:

1. Patients not willing to give informed consent
2. Age less than 16 years
3. Patient presenting with conditions mimicking pilonidal sinus
4. Diabetes mellitus, renal failure, immunosuppression e.g. were excluded

   -

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Superiority of Limberg Flap in Recurrent Pilonidal Sinus Disease | January 2009 to December 2013, Patients were invited for control 1 month, 3 months, 6 months, 1 year intervals
  Superiority as measured by rates of recurrence and complication, length of hospital stay, return work, VAS skore, patient satisfaction and complet healing duration.

REFERENCES:
- [Derived] Bali I, Aziret M, Sozen S, Emir S, Erdem H, Cetinkunar S, Irkorucu O. Effectiveness of Limberg and Karydakis flap in recurrent pilonidal sinus disease. Clinics (Sao Paulo). 2015 May;70(5):350-5. doi: 10.6061/clinics/2015(05)08. Epub 2015 May 1. PMID 26039952